CLINICAL TRIAL: NCT01324388
Title: Pharmacokinetic and Pharmacodynamic Effect of LY2189265 on Lisinopril in Subjects With Hypertension and Metoprolol in Healthy Subjects
Brief Title: A Study of the Effect of LY2189265 on Two Blood Pressure Drugs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11552; H9X-MC-GBCO (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-03-25; First posted 2011-03-29 (Estimated); Results first posted 2014-10-08 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide; Metoprolol; Lisinopril

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- LY2189265 + Lisinopril (Experimental): LY2189265 (dulaglutide): 1.5 milligrams (mg), subcutaneous (SC), on Days 1, 8, 15, and 22 of Part 1 of the study.
  Lisinopril: Dose as prescribed by participant's established course of therapy, oral, daily dosing throughout Part 1 of the study.
  Interventions: Biological: LY2189265; Drug: Lisinopril
- Placebo + Lisinopril (Placebo Comparator): Placebo: 1.5 milligrams (mg), subcutaneous (SC), on Days 1, 8, 15, and 22 of Part 1 of the study.
  Lisinopril: Dose as prescribed by participant's established course of therapy, oral, daily dosing throughout Part 1 of the study.
  Interventions: Drug: Lisinopril; Drug: Placebo
- LY2189265 (Treatment 1)/Metoprolol + LY2189265 (Treatment 2) (Experimental): LY2189265 (dulaglutide): 1.5 milligrams (mg), subcutaneous (SC), on Day 1 of Treatment 1 and on Day 5 of Treatment 2 in Part 2 of the study.
  Metoprolol: 100 mg, oral, on Days 1 through 7 of Treatment 2 in Part 2 of the study.
  There was a washout period of at least 21 days between the LY2189265 and metoprolol doses of each treatment period (Day 1 of Treatment 1 to Day 1 of Treatment 2 in Part 2 of the study).
  Interventions: Biological: LY2189265; Drug: Metoprolol
- Metoprolol + LY2189265 (Treatment 2)/LY2189265 (Treatment 1) (Experimental): LY2189265 (dulaglutide): 1.5 milligrams (mg), subcutaneous (SC), on Day 5 of Treatment 2 and on Day 1 of Treatment 1 in Part 2 of the study.
  Metoprolol: 100 mg, oral, on Days 1 through 7 of Treatment 2 in Part 2 of the study.
  There was a washout period of at least 21 days between the LY2189265 and metoprolol doses of each treatment period (Day 7 of Treatment 2 to Day 1 of Treatment 1 in Part 2 of the study).
  Interventions: Biological: LY2189265; Drug: Metoprolol

INTERVENTIONS:
Biological: LY2189265 — Administered subcutaneously
  Other Names: dulaglutide
  Arms: LY2189265 (Treatment 1)/Metoprolol + LY2189265 (Treatment 2); LY2189265 + Lisinopril; Metoprolol + LY2189265 (Treatment 2)/LY2189265 (Treatment 1)
Drug: Metoprolol — Administered orally
  Arms: LY2189265 (Treatment 1)/Metoprolol + LY2189265 (Treatment 2); Metoprolol + LY2189265 (Treatment 2)/LY2189265 (Treatment 1)
Drug: Lisinopril — Administered orally
  Arms: LY2189265 + Lisinopril; Placebo + Lisinopril
Drug: Placebo — Administered subcutaneously
  Arms: Placebo + Lisinopril

SUMMARY:
The purpose of this study is twofold:

1. To evaluate the effect of LY2189265 on how the body absorbs a blood pressure lowering drug (lisinopril) in participants with high blood pressure who are currently taking lisinopril.
2. To evaluate the effect of LY2189265 on heart rate and blood pressure in healthy volunteers when taken with a Beta-blocker drug (metoprolol).

In Part 1, participants will receive four weekly injections of LY2189265 with continued use of normal lisinopril therapy.

Part 2 is a cross-over study design. Participants will receive a single injection of LY2189265 in one period, and seven daily doses of metoprolol and a single injection of LY2189265 in another period.

ELIGIBILITY:
Inclusion Criteria:

* Male participants: agree to use a reliable method of birth control during the study and for 3 months following the last dose of the investigational product
* Female participants: women not of child-bearing potential due to menopause or surgical sterilization (at least 6 weeks post surgical bilateral oophorectomy, hysterectomy or tubal ligation) confirmed by medical history
* Have a body mass index (BMI) of 18.5 to 40.0 kilograms/square meter (kg/m^2), inclusive at the time of screening
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have venous access sufficient to allow for blood sampling as per the protocol
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study restrictions
* Have given written informed consent on an informed consent form (ICF) approved by Lilly and the corresponding ethics committee (EC) or ethical review board (ERB) governing the site

Part 1 only:

* Have controlled mild to moderate hypertension (supine blood pressure [BP] less than or equal to 140/90 millimeter of mercury (mm Hg) at screening, or results with acceptable deviations that are judged not to be clinically significant by the investigator).
* Males and females with stable medical problems (including Type 2 Diabetes Mellitus [T2DM]) that, in the investigator's opinion, will not significantly alter the disposition of the drug, will not place the participant at increased risk by participating in the study, and will not interfere with interpretation of the data may be included
* Have been on oral antihypertensive medication (lisinopril daily [QD]) for at least 3 months prior to screening, have been on a stable dose for at least 1 month prior to screening, and are, in the investigator's opinion, able to safely adhere to a QD morning dosing regimen. Additional medication may be permitted as indicated

T2DM Participants (Part 1 only):

* Have T2DM controlled with diet or exercise alone or stable on a single oral agent antihyperglycemic medication (metformin, sulfonylureas, repaglinide, nateglinide, acarbose [or other disaccharidase inhibitors] or thiazolidinediones) for at least 3 weeks (3 months for thiazolidinediones) prior to admission
* Have a hemoglobin A1c (HbA1c) value of 6.0% to 9.5% at screening or within 4 weeks prior to screening
* Clinical laboratory test results within normal range or deemed clinically insignificant by the investigator. Abnormalities of serum glucose, serum lipids, urinary glucose, and urinary protein consistent with T2DM are acceptable

Part 2 only:

• Are overtly healthy, as determined by medical history and physical examination

Exclusion Criteria:

* Are currently enrolled in, have completed or discontinued within the last 30 days from, a clinical trial involving an investigational product; or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies to Glucagon-like peptide-1 (GLP-1)-related compounds, including LY2189265, or any components of the formulation
* Are participants who have previously completed or withdrawn from this study, or have taken part in any other study investigating LY2189265 or GLP-1-related compounds within the last 3 months
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have a history or presence of gastrointestinal disorder (including pancreatitis [history of chronic pancreatitis or idiopathic acute pancreatitis] or gall bladder disease) or gastrointestinal disease that impacts gastric emptying (GE) (e.g. gastric bypass surgery, pyloric stenosis) or could be aggravated by GLP-1 analogs (for example; esophageal reflux). Participants having had cholecystectomy (removal of gall bladder) in the past with no further sequelae, may be included in the study at the discretion of the screening physician
* Have a history or presence of thyroid disease, unless have been on a stable dose of thyroxine replacement therapy for at least 1 month
* Show history or evidence of significant active neuropsychiatric disease
* Have personal or family history of medullary thyroid cancer (MTC) or a genetic condition that predisposes to MTC
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Intend to start new concomitant medication during the study, including over-the-counter and herbal medication, use drugs that directly reduce gastrointestinal motility or who regularly use systemic corticosteroids, or potent, inhaled, or intranasal steroids known to have a high rate of systemic absorption
* Have donated more than 500 milliliters (mL) of blood within the month prior to screening
* Have a nondominant arm circumference of greater than 42 centimeters (cm)
* Have an average weekly alcohol intake that exceeds 21 units per week (males up to age 65) and 14 units per week (males over 65 and females), or are unwilling to stop alcohol consumption from 48 hours before each admission until discharge from the unit, and to limit alcohol intake to a maximum of 2 units/day on all other days from screening through 48 hours prior to the follow-up visit. (1 unit = 12 ounces [oz] or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* Are participants who, in the opinion of the investigator, are in any way unsuitable to participate in the study

Part 1 only:

• Have any medical conditions, medical history or are taking any medication which are contraindicated within the lisinopril product information leaflet

Part 2 only:

* Intend to use over-the-counter medication (with the exception of paracetamol and/or antacids) within 7 days prior to dosing or prescription medication (with the exception of vitamin/mineral supplements and/or hormone replacement therapy and/or thyroid replacement therapy) within 14 days prior to dosing of the investigational product
* Have any medical conditions, medical history or are taking any medication which are contraindicated within the metoprolol product information leaflet

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: LY2189265 + Lisinopril: LY2189265 (dulaglutide): 1.5 milligrams (mg), subcutaneous (SC), on Days 1, 8, 15, and 22 of Part 1 of the study.
  Lisinopril: Dose as prescribed by participant's established course of therapy, oral, daily dosing throughout Part 1 of the study.
- Part 1: Placebo + Lisinopril: Placebo: 1.5 milligrams (mg), subcutaneous (SC), on Days 1, 8, 15, and 22 of Part 1 of the study.
  Lisinopril: Dose as prescribed by participant's established course of therapy, oral, daily dosing throughout Part 1 of the study.
- Part 2: LY2189265 First, Then LY2189265 + Metoprolol: LY2189265 (dulaglutide): 1.5 milligrams (mg), subcutaneous (SC), on Day 1 of Treatment 1 and on Day 5 of Treatment 2 in Part 2 of the study.
  Metoprolol: 100 mg, oral, on Days 1 through 7 of Treatment 2 in Part 2 of the study.
  There was a washout period of at least 21 days between the LY2189265 and metoprolol doses of each treatment period (Day 1 of Treatment 1 to Day 1 of Treatment 2 in Part 2 of the study).
- Part 2: LY2189265 + Metoprolol First, Then LY2189265: LY2189265 (dulaglutide): 1.5 milligrams (mg), subcutaneous (SC), on Day 5 of Treatment 2 and on Day 1 of Treatment 1 in Part 2 of the study.
  Metoprolol: 100 mg, oral, on Days 1 through 7 of Treatment 1 in Part 2 of the study.
  There was a washout period of at least 21 days between the LY2189265 and metoprolol doses of each treatment period (Day 7 of Treatment 2 to Day 1 of Treatment 1 in Part 2 of the study).
Period: Part 1 of Study
Arm/Group | Part 1: LY2189265 + Lisinopril | Part 1: Placebo + Lisinopril | Part 2: LY2189265 First, Then LY2189265 + Metoprolol | Part 2: LY2189265 + Metoprolol First, Then LY2189265
Started | 23 | 8 | 0 | 0
Received at Least 1 Dose | 23 | 8 | 0 | 0
Completed | 19 | 6 | 0 | 0
Not Completed | 4 | 2 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Period: Part 2 of Study: First Intervention
Arm/Group | Part 1: LY2189265 + Lisinopril | Part 1: Placebo + Lisinopril | Part 2: LY2189265 First, Then LY2189265 + Metoprolol | Part 2: LY2189265 + Metoprolol First, Then LY2189265
Started | 0 | 0 | 10 | 10
Completed | 0 | 0 | 10 | 9
Not Completed | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Period: Part 2: Washout of at Least 21 Days
Arm/Group | Part 1: LY2189265 + Lisinopril | Part 1: Placebo + Lisinopril | Part 2: LY2189265 First, Then LY2189265 + Metoprolol | Part 2: LY2189265 + Metoprolol First, Then LY2189265
Started | 0 | 0 | 10 | 9
Completed | 0 | 0 | 10 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Part 2 of Study: Second Intervention
Arm/Group | Part 1: LY2189265 + Lisinopril | Part 1: Placebo + Lisinopril | Part 2: LY2189265 First, Then LY2189265 + Metoprolol | Part 2: LY2189265 + Metoprolol First, Then LY2189265
Started | 0 | 0 | 10 | 9
Completed | 0 | 0 | 9 | 9
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of study drug (LY2189265, placebo, or metoprolol).
Groups:
- Part 2: LY2189265 + Metoprolol Crossover: Participants received 2 treatments in Part 2 of the study:
  Treatment 1: LY2189265 (dulaglutide): 1.5 milligrams (mg), subcutaneous (SC), on Day 1
  Treatment 2: LY2189265 (dulaglutide): 1.5 milligrams (mg), subcutaneous (SC), on Day 5; Metoprolol: 100 mg, oral, on Days 1 through 7
  Participants were randomized to 1 of 2 treatment sequences in Part 2 of the study:
  Treatment Sequence A: Treatment 1, Treatment 2
  Treatment Sequence B: Treatment 2, Treatment 1
  There was a washout period of at least 21 days between the LY2189265 and metoprolol doses of each treatment period (Day 1 to Day 1 for Treatment Sequence A and Day 7 to Day 1 for Treatment Sequence B).
- Total: Total of all reporting groups
Arm/Group | Part 1: LY2189265 + Lisinopril | Part 1: Placebo + Lisinopril | Part 2: LY2189265 + Metoprolol Crossover | Total
Number analyzed (Participants) | 23 | 8 | 20 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (10.4) | 54.0 (13.0) | 44.6 (16.7) | 51.8 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 1 | 6 | 18
  Male | 12 | 7 | 14 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 23 | 7 | 18 | 48
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 0 | 8 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 2 | 1 | 11
  White | 9 | 5 | 9 | 23
  More than one race | 2 | 1 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 8 | 20 | 51

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics, Area Under the Concentration Curve (AUC) of Lisinopril
Time Frame: Day -1, Day 3, Day 24 of Part 1
Population: Participants who received at least one dose of study drug (LY2189265 or placebo) with evaluable lisinopril AUC data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (nanograms*hours/milliliter)/milligram
Arm/Group | Part 1: LY2189265 + Lisinopril | Part 1: Placebo + Lisinopril
Number analyzed (Participants) | 23 | 8
(nanograms*hours/milliliter)/milligram
  Day -1 (Baseline) | 1580 (55) | 1740 (26)
  Day 3 (n=22, 8) | 1660 (56) | 1720 (28)
  Day 24 (n=18, 6) | 1540 (52) | 1390 (38)

2. Secondary Outcome: Mean, 24-hour Heart Rate (Collected by Ambulatory Blood Pressure Monitoring [ABPM]) in Response to Co-administration of LY2189265 and Lisinopril
Time Frame: Day -1, Day 3, Day 24 of Part 1
Population: Participants who received at least one dose of study drug (LY2189265 or placebo) with evaluable Part 1 ABPM heart rate data.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Part 1: LY2189265 + Lisinopril | Part 1: Placebo + Lisinopril
Number analyzed (Participants) | 22 | 6
beats per minute (bpm)
  Day -1 (Baseline) | 69.8 (8.9) | 68.9 (6.6)
  Day 3 (n=21, 6) | 78.3 (7.9) | 69.3 (9.0)
  Day 24 (n=18, 6) | 77.1 (9.0) | 71.6 (13.5)

3. Secondary Outcome: Mean, 24-hour Blood Pressure (Collected by Ambulatory Blood Pressure Monitoring [ABPM]) in Response to Co-administration of LY2189265 and Lisinopril
Time Frame: Day -1, Day 3, Day 24 of Part 1
Population: Participants who received at least one dose of study drug (LY2189265 or placebo) with evaluable Part 1 ABPM blood pressure data.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mm Hg)
Arm/Group | Part 1: LY2189265 + Lisinopril | Part 1: Placebo + Lisinopril
Number analyzed (Participants) | 22 | 6
millimeter of mercury (mm Hg)
  Systolic, Day -1 (Baseline) | 129.4 (14.1) | 130.1 (14.9)
  Systolic, Day 3 (n=21, 6) | 125.3 (11.5) | 127.1 (13.4)
  Systolic, Day 24 (n=18, 6) | 121.1 (10.3) | 123.8 (16.2)
  Diastolic, Day -1 (Baseline) | 76.9 (8.6) | 74.1 (7.7)
  Diastolic, Day 3 (n=21, 6) | 77.1 (8.3) | 72.6 (5.1)
  Diastolic, Day 24 (n=18, 6) | 73.8 (9.4) | 71.2 (7.8)

4. Secondary Outcome: Pharmacokinetics, Area Under the Concentration Curve (AUC) of Metoprolol When Administered With LY2189265
Time Frame: Day 4 and Day 7 of Treatment 2 in Part 2
Population: Participants who received at least one dose of study drug (LY2189265 or metoprolol) with evaluable Part 2 metoprolol AUC data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*h/mL)
Arm/Group | Part 2: LY2189265 + Metoprolol Crossover
Number analyzed (Participants) | 20
nanograms*hour per milliliter (ng*h/mL)
  Day 4 | 617 (69)
  Day 7 (n=17) | 813 (63)

5. Secondary Outcome: Pharmacokinetics, Maximum Concentration (Cmax) of Metoprolol When Administered With LY2189265
Time Frame: Day 4 and Day 7 of Treatment 2 in Part 2
Population: Participants who received at least one dose of study drug (LY2189265 or metoprolol) with evaluable Part 2 metoprolol Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Part 2: LY2189265 + Metoprolol Crossover
Number analyzed (Participants) | 20
nanograms per milliliter (ng/mL)
  Day 4 | 35.7 (63)
  Day 7 (n=19) | 47.2 (66)

6. Primary Outcome: Pharmacokinetics, Maximum Concentration (Cmax) of Lisinopril
Time Frame: Day -1, Day 3, Day 24 in Part 1
Population: Participants who received at least one dose of study drug (LY2189265 or placebo) with evaluable lisinopril Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (nanograms per milliliter) per milligram
Arm/Group | Part 1: LY2189265 + Lisinopril | Part 1: Placebo + Lisinopril
Number analyzed (Participants) | 23 | 8
(nanograms per milliliter) per milligram
  Day -1 (Baseline) | 122 (56) | 138 (22)
  Day 3 (n=22, 8) | 114 (55) | 138 (25)
  Day 24 (n=18, 6) | 115 (49) | 110 (39)

7. Primary Outcome: Mean, 24-hour Heart Rate (Collected by Ambulatory Blood Pressure Monitoring [ABPM]) in Response to Co-administration of LY2189265 and Metoprolol
Time Frame: Day -1, Day 4, Day 7 of Treatment 2 in Part 2
Population: Participants who received at least one dose of study drug (LY2189265 or metoprolol) with evaluable Part 2 ABPM heart rate data.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Groups:
- Part 2: LY2189265 + Metoprolol (Treatment 2): Participants received 2 treatments in Part 2 of the study:
  Treatment 1: LY2189265 (dulaglutide): 1.5 milligrams (mg), subcutaneous (SC), on Day 1
  Treatment 2: LY2189265 (dulaglutide): 1.5 milligrams (mg), subcutaneous (SC), on Day 5; Metoprolol: 100 mg, oral, on Days 1 through 7
  Participants were randomized to 1 of 2 treatment sequences in Part 2 of the study:
  Treatment Sequence A: Treatment 1, Treatment 2
  Treatment Sequence B: Treatment 2, Treatment 1
  There was a washout period of at least 21 days between the LY2189265 and metoprolol doses of each treatment period (Day 1 to Day 1 for Treatment Sequence A and Day 7 to Day 1 for Treatment Sequence B).
Arm/Group | Part 2: LY2189265 + Metoprolol (Treatment 2)
Number analyzed (Participants) | 19
beats per minute (bpm)
  Day -1 (Baseline) | 63.7 (9.6)
  Day 4 (n=18) | 55.8 (9.4)
  Day 7 | 69.4 (9.0)

8. Primary Outcome: Mean, 24-hour Blood Pressure (Collected by Ambulatory Blood Pressure Monitoring [ABPM]) in Response to Co-administration of LY2189265 and Metoprolol
Time Frame: Day -1, Day 4, Day 7 of Treatment 2 in Part 2
Population: Participants who received at least one dose of study drug (LY2189265 or metoprolol) with evaluable Part 2 ABPM blood pressure data.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mm Hg)
Groups:
- Part 2: LY2189265 + Metoprolol (Treatment 2): Participants received 2 treatments in Part 2 of the study:
  Treatment 1: LY2189265 (dulaglutide): 1.5 milligrams (mg), subcutaneous (SC), on Day 1
  Treatment 2: LY2189265 (dulaglutide): 1.5 milligrams (mg), subcutaneous (SC), on Day 5 ; Metoprolol: 100 mg, oral, on Days 1 through 7
  Participants were randomized to 1 of 2 treatment sequences in Part 2 of the study:
  Treatment Sequence A: Treatment 1, Treatment 2
  Treatment Sequence B: Treatment 2, Treatment 1
  There was a washout period of at least 21 days between the LY2189265 and metoprolol doses of each treatment period (Day 1 to Day 1 for Treatment Sequence A and Day 7 to Day 1 for Treatment Sequence B).
Arm/Group | Part 2: LY2189265 + Metoprolol (Treatment 2)
Number analyzed (Participants) | 19
millimeter of mercury (mm Hg)
  Systolic, Day -1 (Baseline) | 123.0 (11.4)
  Systolic, Day 4 (n=18) | 115.4 (11.7)
  Systolic, Day 7 | 116.2 (10.4)
  Diastolic, Day -1 (Baseline) | 72.8 (7.3)
  Diastolic, Day 4 (n=18) | 67.2 (7.5)
  Diastolic, Day 7 | 71.8 (6.4)

ADVERSE EVENTS:
Groups:
- Part 2: LY2189265: LY2189265 (dulaglutide): 1.5 milligrams (mg), subcutaneous (SC), on Day 1 of Treatment 1 in Part 2 of the study.
  Time frame: Treatment 1
- Part 2: Metoprolol: Metoprolol: 100 milligrams (mg), oral, on Days 1 through 4 of Treatment 2 in Part 2 of the study.
  Time frame: Days 1 to 4 of Treatment 2
- Part 2: LY2189265 + Metoprolol: LY2189265 (dulaglutide): 1.5 milligrams (mg), subcutaneous (SC), on Day 5 of Treatment 2 in Part 2 of the study.
  Metoprolol: 100 mg, oral, on Days 5 through 7 of Treatment 2 in Part 2 of the study.
  Time frame: Day 5 to end of Treatment 2
Arm/Group | Part 1: LY2189265 + Lisinopril | Part 1: Placebo + Lisinopril | Part 2: LY2189265 | Part 2: Metoprolol | Part 2: LY2189265 + Metoprolol
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/8 | 0/19 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 13/23 | 1/8 | 7/19 | 4/20 | 13/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: LY2189265 + Lisinopril (N=23) | Part 1: Placebo + Lisinopril (N=8) | Part 2: LY2189265 (N=19) | Part 2: Metoprolol (N=20) | Part 2: LY2189265 + Metoprolol (N=19)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 5 (8) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 0 (0) | 5 (5) | 0 (0) | 5 (6)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Device failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural site reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 0 (0) | 6 (6) | 0 (0) | 7 (7)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days